CLINICAL TRIAL: NCT01460056
Title: e-STEPS: Endotoxin-Associated Sterile Peritonitis Observational Study
Acronym: e-STEPS
Status: Completed | Type: Observational
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: M-11378-001
Record Dates: First submitted 2011-10-24; First posted 2011-10-26 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Endotoxin-associated Sterile Peritonitis
Keywords: peritoneal dialysis; endotoxin-associated sterile peritonitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Peritoneal dialysis

SUMMARY:
This observational retrospective healthcare medical record review study is to evaluate and differentiate the clinical characteristics and outcomes in peritoneal dialysis (PD) patients with either endotoxin-associated sterile peritonitis (e-SP), bacterial peritonitis (BP) or no peritonitis (NoP) over a 12-15 month period from dialysis clinics in The Netherlands, Germany, Hungary, Portugal, and the United Kingdom (UK).

The primary study objectives are to:

* Describe changes in the peritoneal membrane function and clinical outcomes over time between e-SP, BP and NoP PD patients.
* Describe and differentiate clinical characteristics during the acute clinical presentation of e-SP and BP.

The secondary study objective is to:

- Generate a dataset that will facilitate post hoc exploratory hypothesis-generation related to clinical and resource utilisation (RU) outcomes in association with e-SP.

DETAILED DESCRIPTION:
e-STEPS is an observational, non-interventional, retrospective review study of healthcare medical records conducted in PD units at approximately 12 sites in The Netherlands, Germany, Hungary, Portugal, and the UK. There will be no study drug or any other medical intervention involved. Furthermore, no patient-identifying information will be transferred to the Study Coordinating Centre (SCC) or the sponsor. Medical records of cases with e-SP, BP and NoP who meet the proposed study selection criteria will be selected from approximately 12 study sites identified across the 5 European countries.

Each case identified by site study staff as potentially eligible for enrollment into the study will be entered into the case disposition log (CDL) and will be assigned a unique site-specific study identification number. These cases will be considered the study sampling frame. The SCC will select a preliminary target cohort of subjects from the sampling frame by selecting all e-SP cases and undertaking a random sample of NoP and BP cases within site to ensure 1:1:1 enrollment ratio between the 3 study groups. In the event that a sampling frame at a given site contains less NoP or BP cases when compared to e-SP cases, all NoP or BP cases will be selected for enrollment into the study and additional cases will be randomly selected from another site within the country to make up for the deficit if sampling frames allow. Sampling within site or alternatively within country ensures that NoP cases are matched to e-SP cases by lot of recalled PD solution. Cases within The Netherlands, Portugal and the UK all used the same recalled lot of PD solutions. Therefore, if within site and within country sampling cannot be achieved, across country sampling can be undertaken in these 3 countries. If it is determined that all e-SP and NoP cases in the sampling frame were on CAPD at the time of the index event, any BP cases identified in the sampling frame on APD at the time of index event may be excluded from the selection process (may not be selected to comprise the preliminary target cohort) and would therefore not be enrolled into the study.

Local site study staff will review the medical records of the cases included in the preliminary target cohort to confirm eligibility. Those cases meeting the eligibility criteria will comprise the final study cohort and will be enrolled into the study as subjects.

Pseudonymised data from the subjects' medical records will be abstracted by local site study staff and entered at the site into the secured pass-word protected electronic data capture (EDC) system. No patient-identifying information will be available to non-site staff; (i.e., representatives of the SCC and the study sponsor). Over the course of the study, as data are entered, the case status page within the EDC system will automatically update the study disposition of each case. As the data will be automatically quality controlled at the point of data entry into the EDC system on the basis of programmed validation rules for each of the study variables, quality control and query resolution can be managed remotely. Therefore, site data monitoring visits by the SCC are not envisioned. No patient-identifying information will be entered into the EDC system; as such, neither the SCC nor the study sponsor will be able to identify subjects as actual patients.

ELIGIBILITY:
1. Endotoxin-associated peritonitis (e-SP) subgroup:

   1.1. Inclusion Criteria:
   * On continuous ambulatory peritoneal dialysis (CAPD) or automated peritoneal dialysis (APD) at time of index event.
   * Used 1 of 3 Baxter PD solutions recalled lots (Nutrineal 10G12G44, Nutrineal 10I13G42, or Dianeal 10I20G44) between 1 August 2010 and 31 December 2010.
   * Has a documented diagnosis of e-SP (index event) between 1 August 2010 and 31 December 2010, defined as meeting 1 of the 2 criteria listed below:
   * Cloudy PD effluent with an increased peritoneal leukocyte count >100 mm3 and a negative bacterial culture; or
   * Cloudy PD effluent which resolves without the use of antibiotics and with the discontinuation of the Baxter PD solutions recalled lot within 24 hours.
   * Aged 18 years or older at time of index event.

   1.2. Exclusion Criteria:
   * Participation in an interventional clinical study (i.e., therapy or dietary interventions) during the applicable study period (from index event to 12-15 months post index event).
   * Had a diagnosis of fungal peritonitis at the index event.
   * Received antibiotics for the treatment of other infectious ailments within 1 week prior to the e-SP index event.
   * Received antibiotics for the treatment of peritonitis (index event) prior to the collection of cloudy PD effluent for cell count and cultures.
   * Had a diagnosis of bacterial peritonitis (BP) within 3 months prior to the e-SP index event.
   * Pregnancy during the applicable study period (from index event to 12-15 months post index event).
2. Bacterial peritonitis (BP) subgroup

   2.1. Inclusion criteria
   * On CAPD or APD at time of index event.
   * Used Baxter's PD solutions lots manufactured by Baxter (Dianeal, Extraneal, Nutrineal in Viaflex containers) between 1 December 2008 and 30 November 2010.
   * Had a documented diagnosis of BP (index event), between 1 December 2008 and 31 December 2010, defined as meeting the 2 criteria listed below:

     * Cloudy peritoneal dialysis (PD) effluent with an increased peritoneal leukocyte count >100 mm3;
     * Positive bacterial culture with a causative organism(s).
   * Aged 18 year or older at time of index event.

   2.2. Exclusion criteria
   * Participation in an interventional clinical study (i.e., therapy or dietary interventions) during the applicable study period (from index event to 12-15 months post index event).
   * Had a diagnosis of e-SP between 1 August 2010 and 31 December 2010.
   * Had a diagnosis of fungal peritonitis at the index event.
   * Pregnancy during the applicable study period (from index event to 12-15 months post index event).
3. No peritonitis (NoP) subgroup

3.1. Inclusion criteria

* On CAPD or APD at time of index event.
* Used 1 of 3 Baxter PD solution recalled lots (Nutrineal 10G12G44, Nutrineal 10I13G42, or Dianeal 10I20G44) between 1 August 2010 and 31 December 2010.
* Aged 18 year or older at time of index event.

3.2. Exclusion criteria

* Had a documented diagnosis of any type of peritonitis between 1 August 2010 and 31 December 2010.
* Participation in an interventional clinical study (i.e., therapy or dietary interventions) during the applicable study period (from index event to 12-15 months post index event).
* Pregnancy during the applicable study period (from index event to 12-15 months post index event).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study subjects will be incident cases of endotoxin-associated peritonitis (e-SP) and bacterial peritonitis (BP) and no peritonitis (NoP) who meet all of the study eligibility criteria during the study eligibility period.
Sampling Method: Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Describe changes in the peritoneal membrane function and clinical outcomes over time between endotoxin associated peritonitis (e-SP), bacterial peritonitis (BP) and no peritonitis (NoP) peritoneal dialysis (PD) patients. | Data will be analysed at 4 time points: baseline, index event, 6±3 months post date of index event, and 12±3 months post date of index event.
  Data including but not limited to demographics, comorbidities, clinical characteristics and outcomes, blood and urine laboratory studies, adequacy and peritoneal membrane function tests, PD prescriptions, empiric antibiotic usage, hospitalisations, outpatient visits, and accident and emergency visits will be collected (retropspective).

CONTACTS AND LOCATIONS:
Overall Officials: Cory Sise, MD, Study Director — Baxter Healthcare Corporation
Locations (12):
- Germany (3):
  - Dialysepraxis Dessau, Dessau
  - Dialysezentrum Würzburg, Würzburg
  - Dialysezentrum Zwickau, Zwickau
- Hungary (3):
  - B.Braun Avitum Zrt. 11 . sz. Dialízisközpont, Győr
  - B.Braun Avitum Zrt. 06 . sz. Dialízisközpont, Szombathely
  - B.Braun Avitum Zrt. 03 . sz. Dialízisközpont, Veszprém
- Netherlands (3):
  - Catharina ziekenhuis, Eindhoven
  - Medisch centrum Haaglanden, The Hague
  - Zaans Medisch Centrum, Zaandam
- Portugal (2):
  - Hospital Évora, Evora
  - Hospital Sao Joao, Porto
- Derriford Hospital, Plymouth, United Kingdom